CLINICAL TRIAL: NCT00531713
Title: Effect of T4-T3 Combination Therapy Versus T4 Monotherapy in Patients With Hypothyroidism,a Double Blind Randomized Cross-Over Study.
Brief Title: Effect of T4-T3 Combination Therapy Versus T4 Monotherapy in Patients With Hypothyroidism
Acronym: T4-T3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: T4-T3 hypothyreose; KA 02022ms
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2007-09-19 (Estimated); Status verified 2007-09

CONDITIONS: Quality of Life; Depression
Keywords: hypothyroidism, quality og life, depression
MeSH Terms: conditions — Depression; Hypothyroidism | interventions — Triiodothyronine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Usual T4 dose is given
- 2 (Active Comparator): 20 microgram of T3 is given and 50 microgram of T4 is withdrawn
  Interventions: Drug: Triiodothyronine

INTERVENTIONS:
Drug: Triiodothyronine — 50 microgram of the usual T4 is withdrawn and the patients is given 20 microgram of T3
  Arms: 2

SUMMARY:
To compare the effect of T4-T3 combination therapy versus T4 monotherapy in patients with autoimmune hypothyroidism, on stable T4-substitution therapy

DETAILED DESCRIPTION:
double blind randomized cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* Hypothyroidism, S-TSH> 20 at diagnosis,Anti-TPO >300 Normal TSH (0,4-4,0) for 6 months.

Exclusion Criteria:

* <18 år
* >75 år
* pregnant women
* Thyroid cancer
* T3 treatment
* Post-partum thyroiditis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2003-04; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Selv-rating scales: SF-36, SCL -90-R, BDI | 3 month treating

SECONDARY OUTCOMES:
BMI, bioimpedance | 3 month treament

CONTACTS AND LOCATIONS:
Overall Officials: Birte Nygaard, Principal Investigator — Herlev Trials
Locations (1):
- Dept of endocrinology , Herlev Hospital, Herlev, Herlev, Denmark